CLINICAL TRIAL: NCT00645450
Title: PTSD Symptom Reduction by Propranolol Given After Memory Activation
Brief Title: PTSD Symptom Reduction by Propranolol Given After Trauma Memory Activation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting subjects and loss of study physician for new job
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBA-013-07S
Record Dates: First submitted 2008-03-19; First posted 2008-03-27 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Posttraumatic Stress Disorders
Keywords: Stress; Posttraumatic; PTSD; Propranolol; Treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Experimental): Weekly doses of short and long acting propranolol following recollection of traumatic memory
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): Weekly doses of placebo following recollection of traumatic memory
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Weekly doses of short and long acting propranolol (Inderal, Inderal LA, Hemangeol, Inderal XL) following recollection of traumatic memory
  Other Names: Inderal, Inderal LA, Hemangeol, Inderal XL
  Arms: Propranolol
Drug: Placebo — Weekly doses of placebo (inactive pill) following recollection of traumatic memory
  Other Names: Inactive pill
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled clinical trial of propranolol combined with trauma memory reactivation, to determination if this approach is effective in treating PTSD symptoms. Participants will include male and female combat Veterans of the Afghanistan and Iraqi wars meeting DSM-IV criteria for chronic PTSD, recruited locally from the Manchester VAMC Mental Hygiene Clinic or through advertising. The presence of PTSD will be assessed using the CAPS. Participants will be randomly assigned to the propranolol or placebo drug condition. During each of six memory reactivation sessions, the participant will meet with a psychiatrist, who will ask the participant to spend ten minutes describing the event that caused their PTSD, and their reactions to it. The interviewer will facilitate this process by asking questions, keeping the participant focused on the traumatic event and encouraging him/her to identify aspects of the traumatic event that continue to provoke emotional distress. The traumatic memory reactivation will be immediately followed by administration of propranolol or placebo. Following the six treatment sessions, script-driven imagery will be used to assess HR, SC, and facial EMG responses to recollections of the traumatic event and PTSD symptoms will be assessed using the CAPS. A previously developed discriminant function will be used to classify each person as a physiologic "responder" or "non-responder." There will also be a 6-month follow-up assessment.

DETAILED DESCRIPTION:
OBJECTIVE: In the first of two preliminary studies, the investigators demonstrated in individuals with chronic PTSD that a single (combined 40 mg short- and 60 mg long-acting) 24-hour oral dose of propranolol, compared to placebo, given immediately following reactivation of the PTSD-related memory of the traumatic event, significantly reduced physiological responses during script-driven imagery of that event measured one week later. These results support blockade of reconsolidation of the traumatic memory, a process that is entirely distinct from extinction. In addition, the investigators found a trend for post-reactivation propranolol to reduce self-reported PTSD symptoms, measured via the Impact of Event Scale-Revised (IES-R). In the second preliminary study, the investigators performed 6 weekly treatments that consisted of the subject describing their PTSD-related traumatic events for approximately 10 minutes followed by 0.67 mg/kg (minimum 40 mg) short-acting propranolol plus 1 mg/kg (minimum 60 mg) long-acting propranolol. The mean Clinician Administered PTSD Scale (CAPS) Total Score following the six treatment sessions was reduced by 44% (p=.02). The proposed work will examine whether repeated treatments may succeed in producing more substantive symptomatic improvement.

RESEARCH PLAN: The study design will be a randomized, double-blind, placebo-controlled, clinical trial. A crossover design is not being proposed because the effect is expected to be neither short-term nor reversible. Rather, at the conclusion of the formal study period, individuals randomized to the placebo condition will be offered an equal number of treatment sessions with propranolol. A placebo control will be used, rather than an active treatment control, because the proposed study will be a "proof of concept" test of post-reactivation pharmacological reduction of traumatic memories. The control (and active) treatments will be structured so as to minimize the chance of extinction. The investigators recognize that eventually this new treatment will need to be tested against established PTSD treatments, including exposure, if its clinical utility is to be established. The investigators regard this as a matter for subsequent studies should the present study yield promising results. However, the investigators do intend to compare the effect size the investigators find for the proposed intervention with published effect sizes for other PTSD psychotherapies.

METHODOLOGY: Participants will include male and female combat Veterans of the Afghanistan and Iraqi wars meeting DSM-IV criteria for chronic PTSD, recruited locally from the Manchester VAMC Mental Hygiene Clinic or through advertising. The presence of PTSD will be assessed using the CAPS. Participants will be randomly assigned to the propranolol or placebo drug condition. During each of six memory reactivation sessions, the participant will meet with a psychiatrist, who will ask the participant to spend ten minutes describing the event that caused their PTSD, and their reactions to it. The interviewer will facilitate this process by asking questions, keeping the participant focused on the traumatic event and encouraging him/her to identify aspects of the traumatic event that continue to provoke emotional distress. The traumatic memory reactivation will be immediately followed by administration of propranolol or placebo. Following the six treatment sessions, script-driven imagery will be used to assess HR, SC, and facial EMG responses to recollections of the traumatic event and PTSD symptoms will be assessed using the CAPS. A previously developed discriminant function will be used to classify each person as a physiologic "responder" or "non-responder." There will also be a 6-month follow-up assessment.

CLINICAL RELEVANCE: The mechanism of memory reconsolidation offers the possibility that cellular plasticity can be capitalized on to reverse the neuroanatomical and neurophysiological underpinnings of traumatic memories. The possibility that a traumatic memory could be significantly weakened by an intervention as simple as the post-reactivation administration of a widely used and safe medication has profound implications for the treatment of PTSD.

ELIGIBILITY:
Inclusion Criteria:

OEF/OIF veteran diagnosed with combat related posttraumatic stress disorder

Exclusion Criteria:

1. Not diagnosed with current, chronic PTSD
2. Current PTSD related to a traumatic event other than the event being treated
3. Age>65.
4. Systolic blood pressure <100 mm HG or resting HR less than 60 BPM.
5. Medical condition that contraindicates the administration of propranolol, e.g. history of congestive heart failure, heart block, insulin-requiring diabetes, chronic bronchitis, emphysema, or asthma. With regard to asthma, because many persons who say they have had an asthma attack, especially as a child, may only have had hay fever, another allergy, or another non-asthmatic episode, a blanket exclusion criteria may be overly restrictive. Therefore asthma attacks will only be exclusionary if they a) occurred within the past 10 years, b) occurred at any time in life if induced by a beta-blocker, or c) are currently being treated, regardless of the date of last occurrence. Cardiological consultation will be obtained as necessary;
6. Previous adverse reaction to, or non-compliance with a beta-blocker.
7. Current use of medication that may involve potentially dangerous interactions with propranolol, including, other beta-blockers, antiarrhythmics, calcium channel blockers, and potent P450 2D6 inhibitors, e.g., fluoxetine, paroxetine, micnazole, sulconazole, metaclopramide, quinidine, ticlopidine, and ritnavir.
8. Presence of drugs of abuse, viz., opiates, marijuana, cocaine, or amphetamines, as determined by urine testing.
9. Pregnancy (in women of child- bearing potential, a pregnancy test will be performed) or breast feeding.
10. Contraindicating psychiatric condition, e.g., current psychotic, bipolar, melancholic, or substance dependence or abuse disorder.
11. Initiation of, or change in, psychotropic medication within the previous two months. For subjects receiving stable doses of pharmacotherapy, they and their providers will be asked not to change the regimen except in clinically urgent circumstances. If this becomes necessary, a decision will be made on a case-by-case basis whether to retain the subject in the study or terminate participation.
12. Current participation in any psychotherapy (other than supportive). Subjects will be asked not to initiate psychotherapy during the course of the proposed study except in clinically urgent circumstances; if this becomes necessary, a decision will be made on a case-by-case basis whether to retain the subject in the study or terminate participation.
13. Inability to understand the study's procedures, risks, and side effects, or to otherwise give informed consent for participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott P Orr, PhD, Principal Investigator — VA Medical Center, Manchester
Locations (1):
- VA Medical Center, Manchester, Manchester, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
Study terminated early.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propranolol | Placebo
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants included combat Veterans of Afghanistan and Iraqi wars.
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol | Placebo | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (4.62) | 25.5 (.71) | 27 (3.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 4 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptom Severity as Measured by Clinician-Administered PTSD Scale (CAPS)
Description: CAPS scale measures intensity and frequency of each symptom separately on a 5 point Likert scale ranging from zero to four. The total CAPS symptom severity score ranges from 0-136, with higher scores indicating greater PTSD symptoms severity
Time Frame: 3 years
Population: Data does not include subjects who consented but withdrew prior to receiving study intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 3 | 2
score on a scale | 2.60 (1.27) | 2.19 (3.10)

ADVERSE EVENTS:
Arm/Group | Propranolol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol (N=5) | Placebo (N=4)
Incorrect dosage (Cardiac disorders) | 1 (1) | 0 (0) — Incorrect dosage of Propranolol no adverse medical effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No